CLINICAL TRIAL: NCT01137617
Title: Effect of Spinal Cord Stimulation on Pain Thresholds and Sensory Perception in Chronic Pain Patients.
Acronym: SCS
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jianren Mao, MD, PhD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2010P 000425
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Chronic Pain
Keywords: spinal cord stimualtor
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to better understand how the Spinal Cord Stimulator works in relieving chronic pain.

The investigators are asking subject to take part in this study because who are chronic pain patients who already have a Spinal Cord Stimulator (SCS) in place.

The investigators hypothesize that chronic pain patients will have higher heat pain threshold and heat pain tolerance over the painful areas with the SCS on.

QST (Quantitative Sensory Testing, a heat/cold simulation test) might be an objective helpful tool for prudent patient selection for an expensive and invasive procedure for future SCS placement.

DETAILED DESCRIPTION:
Sixty subjects who already have an implanted SCS device for pain management at the MGH Center for Pain Medicine and other Partners affiliated pain centers will be enrolled.

Inclusion Criteria:

1. Subject is 18 years or older.
2. Subject has an SCS device implanted for at least one month for pain control. This requirement is set to ensure that the subject becomes familiarized with the therapy and has recovered from the surgical implantation of the SCS device.

Exclusion Criteria:

1. Subject has neurological disease or a condition causing sensory deficit to the painful area.
2. Subject had recent therapy that may influence QST results, e.g., neuroablative procedure within two-months.
3. Subjects who are unable to travel to the study center.

It will be a one time outpatient visit study, which will include the following:

1. Brief pain history and Neurological examination

   * Medical History (including medication use);
   * Pain location, intensity, character and if known, etiology, duration;
   * Maps of pain locations and paresthesia locations;
   * Sensory neurological examination (e.g., alcohol swab, cotton swab, pinprick and vibration);
   * A check on routine vital signs (blood pressure, pulse, pulse oximetry).
2. QST will include the following:

   * Warm sensation, heat pain threshold, heat pain tolerance and wind-up. A cut-off of 53°C for heat will be preset to avoid tissue damage.
   * QST will be done on two areas; painful area and non-painful area without paresthesia with the SCS turned off.
   * Subject will then turn on SCS and a repeat QST will be performed on the painful and non-painful areas.
   * QST tests will be performed in a quiet room at temperature 25º 2° C. The time and duration of the QST tests will be recorded.

QST will be performed at least 4 hours and no later than 6 hours after the last dose of long acting opioid and after last SCS on time. In this way the investigators will try to avoid recording possible end dose withdrawal and provide sufficient time for the subject to return to baseline for their SCS therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years or older.
* Subject has an SCS device implanted for at least one month for pain control. This requirement is set to ensure that the subject becomes familiarized with the therapy and has recovered from the surgical implantation of the SCS device.

Exclusion Criteria:

* Subject has neurological disease or a condition causing sensory deficit to the painful area.
* Subject had recent therapy that may influence QST results, e.g., neuroablative procedure within two-months.
* Subjects who are unable to travel to the study center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixty subjects who already have an implanted SCS device for pain management at the MGH Center for Pain Medicine and other Partners affiliated pain centers will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2010-06; Primary Completion 2011-08 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Warm Sensation (WS) Threshold- Pain Site | WS threshold is assessed once at Visit 1
  WS threshold is a type of Quantitative Sensory Test (QST). A contact thermode was attached to the subject's painful area that has SCS coverage. The thermode increased by 1°C/sec from a baseline of 32°C. Subjects were instructed to stop stimulation when they first perceived a warm sensation. Subjects performed this test with their SCS off and again with their SCS on.
Heat Pain (HP) Threshold- Pain Site | HP threshold is assessed once at Visit 1
  Heat Pain threshold is a type of QST. A contact thermode was attached to the subject's painful area that has SCS coverage. The thermode increased by 1°C/sec from a baseline of 32°C. Subjects were instructed to stop the stimulation when pain was first detected. Subjects performed this test with their SCS off and again with their SCS on.
Heat Pain Tolerance- Pain Site | Heat Pain Tolerance is assessed once at Visit 1
  Heat Pain threshold is a type of QST. A contact thermode was attached to the subject's painful area that has SCS coverage. The thermode increased by 1°C/sec from a baseline of 32°C. Subjects were instructed to stop the stimulation when pain was no longer tolerable. Subjects performed this test with their SCS off and again with their SCS on.

CONTACTS AND LOCATIONS:
Overall Officials: Shihab Ahmed, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Center for Translational Pain Research, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No